CLINICAL TRIAL: NCT02557945
Title: Gabapentin in Patients at Clinical Risk for Psychosis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Combination of insufficient funding and lack of compelling findings
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Scott Small, Professor of Neurology, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 7165R
Record Dates: First submitted 2015-08-31; First posted 2015-09-23 (Estimated); Results first posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Clinical High Risk for Psychosis
MeSH Terms: interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gabapentin (Experimental): Gabapentin 3600mg PO daily
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator): Matching placebo PO daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — Subjects will be treated with 400mg pills of gabapentin , titrating up to 3600mg per day, or 9 tablets (3 tabs tid)
  Arms: Gabapentin
Drug: Placebo — Subjects will be treated with 400mg pills of placebo, titrating up to 3600mg per day, or 9 tablets (3 tabs tid)
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the effects of the drug gabapentin on brain function thought to be important in the development of schizophrenia. Researchers think that treating a brain region with gabapentin (the hippocampus) may reduce the risk for developing schizophrenia.

DETAILED DESCRIPTION:
Six week, single site, proof-of concept, randomized double-blind placebo-controlled pilot study to examine the effects of moderate dose gabapentin (3600mg) in n= 100 putatively prodromal patients on hippocampal activity.

ELIGIBILITY:
Inclusion Criteria:

1. COPE patient between age of 18-30
2. Capacity to give informed consent
3. Currently using a reliable method of birth control (female) (condom plus spermicide, diaphragm plus spermicide, IUD, birth control pills, norplant, vasectomy in partner)

Exclusion Criteria:

1. Metal implants in body or a history of metal working, or more than one past MRI scan with gadolinium
2. Lifetime diagnosis of asthmatic symptoms within the past 3 years or known sensitivity to contrast agents
3. Lifetime diagnosis of renal failure/disease
4. Acute neurological, neuroendocrine,or medical disorder including renal insufficiency
5. Lifetime diagnosis of hypertension or diabetes
6. Intelligence Quotient (IQ) < 70
7. Acute risk for suicide and/or violence
8. Pregnant, lactating
9. Current abuse of substances (alcohol, cocaine, stimulants, cannabis, opiates, sedative hypnotics)
10. Current use or anticipated need for antipsychotics or mood stabilizers (all antipsychotics, also Depakote, lithium, lamotrigine, pregabalin or any med with a mechanism of action like gabapentin)
11. The Clinical Global Impressions Scale (CGI)-improvement score during study equal to or greater than 6

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2016-06-12 (Actual); Study Completion 2016-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ragy Girgis, M.D., Principal Investigator — NYSPI/Columbia
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 9 individuals signed consent and underwent screening procedures for the study. 6 of the 9 were randomized to receive gabapentin/placebo
Period: Overall Study
Arm/Group | Gabapentin | Placebo
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline population are the individuals who received gabapentin or placebo and underwent MRI procedures
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Placebo | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Left CA1 Cerebral Blood Volume (CBV) (MRI Measure)
Description: Change from 6 week follow up minus baseline of left CA1 CBV (MRI measure) in patients who receive active drug vs. placebo, after 6 weeks of treatment.
Time Frame: 6 weeks
Population: While 6 participants received gabapentin or placebo, 1 participant data was excluded due to low quality of scans. Only 5 participants data were analyzes (2 in gabapentin group, 3 in placebo group)
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 2 | 3
percent change | -0.005 (0.388) | 0.38 (0.317)

2. Secondary Outcome: Change in Positive, Negative, Disorganization, and General Symptoms Over Time as Measured by the Structured Interview for Psychosis-Risk Syndromes (SIPS)/the Scale of Psychosis-Risk Symptoms (SOPS)
Description: Exploratory analyses will be conducted examining the effects of gabapentin on changes in Positive symptoms (P scores), negative symptoms (N scores) and general symptoms (G scores) and disorganization symptoms (D scores) compared to placebo. There are 19 items on the SIPS. Each item is scored 0-6. There are 5 positive symptom items (range=0-30), 6 negative symptom items (range=0-36), 4 disorganization symptom items (range=0-24), and 4 general symptom items (range=0-24). The range of scores is 0-114. A lower score at baseline indicates less symptoms, and therefore a negative change over the 6 week period indicates an improvement, and a positive change indicates worsening of symptoms.
Time Frame: 6 weeks
Population: For general symptom score (G score) and disorganization symptom (D score), 1 participant had missing data and was not included in the data reporting.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 2 | 3
score on a scale
  P score change | -1.5 [-2 to -1] | 0.66 [0 to 2]
  N score change | -1 [-4 to 2] | -1.66 [-5 to 3]
  G score change: number analyzed (Participants) | 2 | 2
  G score change | -1.5 [-2 to -1] | 0.5 [0 to 1]
  D score change: number analyzed (Participants) | 2 | 2
  D score change | 2 [1 to 3] | -2.5 [-5 to 0]

3. Secondary Outcome: Change in Cognitive Function (Hippocampal-dependent Verbal Memory) as Measured by the California Verbal Learning Test-Second Edition (CLVT-II)
Description: Exploratory analyses will be conducted on changes between gabapentin and placebo groups on the California Verbal Learning Test-Second Edition (CLVT-II) measures. The unit measured was 'learning slope', where higher slope indicates better memory and a lower slope indicates poorer memory.
Time Frame: 6 weeks
Measure: Mean (Full Range); unit: Change in raw learning slope
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 2 | 3
Change in raw learning slope | 0.1 [0.1 to 0.1] | -0.3 [-0.6 to 0.2]

ADVERSE EVENTS:
Time Frame: From consent to completion of participation (approximately 42 days)
Arm/Group | Gabapentin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 1/3 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin (N=3) | Placebo (N=3)
paresthesias (Nervous system disorders) | 1 (1) | 0 (0) — mild, transient paresthesias

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes